CLINICAL TRIAL: NCT00636493
Title: A Pilot Study of a Sustained-Release Fluocinolone Implant for Treatment of Retinal Vein Occlusion
Brief Title: Fluocinolone Acetonide Implant for Retinal Vein Occlusion (RVO)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Glenn Jaffe (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor-Investigator, Glenn Jaffe, Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00010864 (3964)
Record Dates: First submitted 2008-02-27; First posted 2008-03-14 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Retinal Vein Occlusion
Keywords: retinal vein occlusion; sustained drug delivery implant; steroid; macular edema
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vein Occlusion Eye (Experimental): Eye with retinal vein occlusion receiving fluocinolone acetonide sustained drug delivery device
  Interventions: Device: fluocinolone acetonide (Retisert Implant)

INTERVENTIONS:
Device: fluocinolone acetonide (Retisert Implant) — sustained release device consisting of 0.59 mg of fluocinolone acetonide
  Other Names: Retisert Implant, Bausch and Lomb, Rochester, NY

SUMMARY:
Purpose: To determine whether a fluocinolone acetonide sustained drug delivery implant is effective in the treatment of retinal vein occlusion that has caused persistent macular edema and decreased visual acuity.

Hypothesis: A fluocinolone acetonide sustained drug delivery implant will be a safe and effective method to treat patients with macular edema and decreased vision from retinal vein occlusion.

DETAILED DESCRIPTION:
Currently there is limited treatment for macular edema and vision loss due to retinal vein occlusion. Case reports have shown some benefit of intravitreal steroid injections in improving vision and reducing macular edema in eyes with retinal vein occlusions.

Recently, a sustained drug release steroid implant has been investigated and FDA approved to treat macular edema in patients with non-infectious uveitis, eye inflammation. This implant is placed through an incision in the eye wall and is designed to deliver a steroid, fluocinolone acetonide, for upto three years. In animal studies there was no detectable steroid seen in the blood stream.

This pilot trial will recruit individuals who have had a retinal vein occlusion in at least one eye. If the macular edema and vision improves with an initial intravitreal injection, the eye will be considered to receive the sustained drug release device. The dosage of fluocinolone acetonide used is 0.59 mg.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to receive an implant if they met all the following criteria:

* A history of retinal vein occlusion that had caused macular edema, based on clinical evaluation and demonstrated on fundus photography, fluorescein angiography, and optical coherence tomography (OCT)
* Macular edema at least one disc area in size that involved the fovea
* Males and non-pregnant females at least 18 years of age
* Intraocular Pressure (IOP) controlled at < 21 mmHg with no more than one topical ocular antihypertensive agent
* Ability and willingness to comply with treatment and follow up process and to understand and sign the informed consent form.
* Initially, patients with vein occlusion were not required to have previous therapy. However, the protocol was subsequently modified to require an intravitreal injection of triamcinolone acetonide > 12 weeks prior to study entry, with an initial decrease in macular edema and improvement in visual acuity and subsequent decline in visual acuity accompanied by increased macular edema. This modification was added to avoid enrolling patients who might have had a long-lasting response to a single intravitreal triamcinolone acetonide injection.

Exclusion Criteria:

* Patients are excluded if they have an allergy to fluocinolone acetonide or any component of the delivery system, a peripheral retinal detachment in the area of implantation, or media opacity precluding evaluation of study eye status.
* Patents with disciform scars of the fovea or atrophic changes of the macula that in the investigator's opinion would preclude benefit from treatment are excluded from the study.
* Female patients who were pregnant or lactating or not taking precautions to avoid pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in visual acuity using Early Treatment Diabetic Retinopathy Study (ETDRS) charts | preoperatively, postoperative day 1, week 1, 1 month, 2 months, 6 months, 9 months, 12 months, then every 13 weeks thereafter for a total of 4 years

SECONDARY OUTCOMES:
Amount of macular edema on optical coherence tomography and color photos | preoperatively, postoperative day 1, week 1, 1 month, 2 months, 6 months, 9 months, 12 months, then every 13 weeks thereafter for a total of 4 years
Elevations in Intraocular Pressure (IOP) requiring anti-glaucoma medication or increase in number of medications required or need for drainage surgery to maintain IOP within clinically satisfactory levels. | preoperatively, postoperative day 1, week 1, 1 month, 2 months, 6 months, 9 months, 12 months, then every 13 weeks thereafter for a total of 4 years
Quality of life scores using the Visual Functioning (VF)-25 and SF-36 surveys | preoperatively, postoperative day 1, week 1, 1 month, 2 months, 6 months, 9 months, 12 months, then every 13 weeks thereafter for a total of 4 years
Ocular adverse events (vitreous hemorrhage, retinal detachment, cataract, endophthalmitis, drug toxicity) | preoperatively, postoperative day 1, week 1, 1 month, 2 months, 6 months, 9 months, 12 months, then every 13 weeks thereafter for a total of 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Jaffe, MD, Principal Investigator — Duke Eye Center, DUMC
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Jaffe GJ, Martin D, Callanan D, Pearson PA, Levy B, Comstock T; Fluocinolone Acetonide Uveitis Study Group. Fluocinolone acetonide implant (Retisert) for noninfectious posterior uveitis: thirty-four-week results of a multicenter randomized clinical study. Ophthalmology. 2006 Jun;113(6):1020-7. doi: 10.1016/j.ophtha.2006.02.021. Epub 2006 May 9. PMID 16690128
- [Background] Jaffe GJ, McCallum RM, Branchaud B, Skalak C, Butuner Z, Ashton P. Long-term follow-up results of a pilot trial of a fluocinolone acetonide implant to treat posterior uveitis. Ophthalmology. 2005 Jul;112(7):1192-8. doi: 10.1016/j.ophtha.2005.03.013. PMID 15921758
- [Background] Jaffe GJ, Ben-Nun J, Guo H, Dunn JP, Ashton P. Fluocinolone acetonide sustained drug delivery device to treat severe uveitis. Ophthalmology. 2000 Nov;107(11):2024-33. doi: 10.1016/s0161-6420(00)00466-8. PMID 11054326